CLINICAL TRIAL: NCT02871726
Title: Transrectal Ultrasound Robot-Assisted Prostate Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00068488
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer Detection; Prostate Biopsy; Prostate Cancer; Transrectal Ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRUS-Robot and TRUS (Experimental): TRUS and TRUS-Robot will be used during prostate biopsy
  Interventions: Device: TRUS-Robot; Other: TRUS biopsy
- Routine TRUS/Fusion biopsy (Active Comparator): Just Uronav will be used during prostate biopsy
  Interventions: Other: TRUS biopsy

INTERVENTIONS:
Device: TRUS-Robot — A robotic device used to hold and manipulate the ultrasound probe during a transrectal prostate biopsy.
  Arms: TRUS-Robot and TRUS
Other: TRUS biopsy — Uronav for prostate biopsy.

SUMMARY:
Prostate cancer (PCa) is the most common non-dermatologic malignancy in U.S. men. Transrectal ultrasound (TRUS)-guided prostate biopsy is a commonly used diagnostic procedure for men with an elevated serum prostate-specific antigen (PSA) level and/or abnormal digital rectal examination (DRE). It is estimated that more than 1 million TRUS-guided prostate biopsies are performed annually in the U.S. alone. However, a freehand TRUS-guided systematic biopsy (SB) procedure has significant limitations. First, freehand biopsy cores are often spatially clustered, rather than uniformly distributed, and do not accurately follow the recommended, sextant template. Second, a freehand TRUS-guided biopsy does not allow precise mapping of the biopsy cores within the prostate. Targeted biopsy (TB) using special devices emerged to help the physicians guide the biopsy using multiparametric MRI (mpMRI). TB cores yield a higher cancer detection rate of clinically significance PCa than SB cores, but TB cores also miss a large number of clinically significant PCa that are detected by SB. Accordingly, TB is commonly performed concurrently with SB (TB+SB procedure).

DETAILED DESCRIPTION:
This study attempts to improve TRUS-guided prostate biopsy by utilizing assistance from a novel robotic TRUS manipulator (TRUS-Robot) developed by our team. The hypothesis of the study is that clinically significant prostate cancer detection rate from the SB cores (at SB or TB+SB) can be improved above that of current devices. The objective of the study is to gain early evidence on the effectiveness of prostate biopsy assisted by the TRUS-Robot vs. a current TB device in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an initial diagnostic biopsy
* Elevated serum PSA (prostate specific antigen> 4 ng/ml) and/or abnormal digital rectal exam

Exclusion Criteria:

* Clinical diagnosis of prostate cancer
* Prior prostate biopsy
* Anal stenosis that prevents TRUS probe insertion
* Inadequate bowel prep
* Unwilling or unable to sign the informed consent

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate of Clinically Significant Prostate Cancer | 5 years
  Number of biopsy patients diagnosed with Gleason score >= 7 over the total number of patients on both arms of the study.
Investigational device serious adverse events | 5 years
  Serious adverse events will be assessed according to 21 Code of Federal Regulations (CFR) Part 812.3(s).
Cancer Detection Rate of Clinically Insignificant Prostate Cancer | 5 years
  Number of biopsy patients diagnosed with Gleason score <= 6 over the total number of patients on both arms of the study.

SECONDARY OUTCOMES:
Needle targeting accuracy | 5 years
  Needle targeting errors will be measured as the distance between the planned core center and the inserted needle axis. Targeting accuracy will be calculated as the average of the needle targeting errors, as usual.
Procedure time | Up to 30 minutes
  The time of the actual biopsy procedure measured in minutes.
Sensitivity of detecting clinically significant prostate cancer at biopsy | 5 years
  Compare biopsy pathology results with gold standard pathology on the subset of patients who follow on to radical prostatectomy. Perform binary tests (True/False x Positive/Negative) and calculate sensitivity.
Specificity of detecting clinically significant prostate cancer at biopsy | 5 years
  Compare biopsy pathology results with gold standard pathology on the subset of patients who follow on to radical prostatectomy. Perform binary tests (True/False x Positive/Negative) and calculate specificity.
Predictive rates of detecting clinically significant prostate cancer at biopsy | 5 years
  Compare biopsy pathology results with gold standard pathology on the subset of patients who follow on to radical prostatectomy. Perform binary tests (True/False x Positive/Negative) and calculate predictive rates.

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, M.D., M.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No